CLINICAL TRIAL: NCT01689142
Title: A 6-Month, Multicenter, Randomized, Open-label, Parallel-group Study Comparing the Efficacy and Safety of a New Formulation of Insulin Glargine and Lantus® Both in Combination With Oral Antihyperglycemic Drug(s) in Japanese Patients With Type 2 Diabetes Mellitus With a 6 Month Safety Extension Period
Brief Title: Comparison of a New Formulation of Insulin Glargine With Lantus® Both in Combination With Oral Antihyperglycemic Drug(s) in Japanese Patients With Type 2 Diabetes Mellitus
Acronym: EDITION JP II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC12512; U1111-1130-3649 (Other: UTN)
Record Dates: First submitted 2012-09-14; First posted 2012-09-21 (Estimated); Last update posted 2014-06-05 (Estimated); Status verified 2014-06

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- New formulation of insulin glargine (Experimental): once daily in the evening on-top of oral antihyperglycemic drug (OADs)
  Interventions: Drug: Insulin glargine new formulation (HOE901)
- Lantus (insulin glargine) (Active Comparator): once daily in the evening on-top of OADs
  Interventions: Drug: Insulin glargine (HOE901)

INTERVENTIONS:
Drug: Insulin glargine new formulation (HOE901) — Pharmaceutical form: solution Route of administration: subcutaneous
  Arms: New formulation of insulin glargine
Drug: Insulin glargine (HOE901) — Pharmaceutical form: solution Route of administration: subcutaneous
  Other Names: Lantus
  Arms: Lantus (insulin glargine)

SUMMARY:
Primary Objective:

To compare the efficacy of a new formulation of insulin glargine and Lantus in terms of change of HbA1c from baseline to endpoint (scheduled at month 6 [week 26]) in japanese patients with type 2 diabetes mellitus.

Secondary Objectives:

To compare a new formulation of insulin glargine and Lantus in terms of change in fasting plasma glucose (FPG), preinjection plasma glucose, 8-point self-measured plasma glucose (SMPG) profile.

To compare a new formulation of insulin glargine and Lantus in terms of occurrence of hypoglycemia

DETAILED DESCRIPTION:
The duration of study will consist of:

* Up to 2-week screening period;
* 6-month open-label comparative efficacy and safety treatment period;
* 6-month open-label comparative safety extension period;
* 4-week post-treatment safety follow-up period

ELIGIBILITY:
Inclusion criteria :

o Patients with type 2 diabetes mellitus diagnosed for at least 1 year at the time of screening visit treated with basal insulin in combination with oral antihyperglycemic drugs (OADs) for at least 6 months before screening visit;

Exclusion criteria:

* Age < 18 years at screening visit;
* BMI(body mass index) ≥ 35 kg/m2 at screening visit;
* HbA1c < 7.0% or > 10% (national glycohemoglobin standardization program [NGSP] value) at screening visit;
* Diabetes other than type 2 diabetes mellitus;
* Patients on self-monitoring of blood glucose less than 6 months before screening visit;
* Patients using pre-mix insulins, insulin detemir at 2 times or more a day, or GLP 1 receptor agonists in the last 3 months before screening visit;
* Patients using mealtime insulin (rapid-acting insulin analogue and short-acting insulin) for more than 10 days in the last 3 months before screening visit;
* Use of insulin pump in the last 6 months before screening visit;
* Initiation of new glucose-lowering medications and/or weight loss drugs in the last 3 months before screening visit;
* Severe hypoglycemia resulting in coma/seizures, and/or hospitalization for diabetic ketoacidosis in the last 6 months before screening visit;
* Unstable proliferative diabetic retinopathy or any other rapidly progressive diabetic retinopathy or macular edema likely to require treatment (eg, laser, surgical treatment or injectable drugs) during the study period.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2012-09; Primary Completion 2013-11 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HbA1c | baseline, 6 months

SECONDARY OUTCOMES:
Percentage of HbA1c responders (HbA1c < 7%; < 6.5%) | up to 6 months
Change from baseline in FPG | baseline, 6 months
Change from baseline in pre-basal insulin injection SMPG | baseline, 6 months
Change from baseline in 8-point SMPG profiles | baseline, 6 months
Change from baseline in 24-hour mean plasma glucose of SMPG profiles (mean of 8-point values) | baseline, 6 months
Change from baseline in variability of plasma glucose profile | baseline, 6 months
Change from baseline in daily basal insulin dose | baseline, 6 months
Number of patients with various types of hypoglycemia events | up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (31):
- Japan (31):
  - Investigational Site Number 392226, Amagasaki-Shi
  - Investigational Site Number 392218, Chigasaki-Shi
  - Investigational Site Number 392212, Chiyoda-Ku
  - Investigational Site Number 392208, Chuoh-Ku
  - Investigational Site Number 392209, Chūōku
  - Investigational Site Number 392210, Chūōku
  - Investigational Site Number 392217, Ebina-Shi
  - Investigational Site Number 392216, Fujisawa-Shi
  - Investigational Site Number 392222, Higashiosaka-Shi
  - Investigational Site Number 392223, Izumisano
  - Investigational Site Number 392215, Kamakura-Shi
  - Investigational Site Number 392225, Kashiwara-Shi
  - Investigational Site Number 392205, Kawagoe-Shi
  - Investigational Site Number 392204, Kawaguchi-Shi
  - Investigational Site Number 392206, Kisarazu-Shi
  - Investigational Site Number 392201, Koriyama-Shi
  - Investigational Site Number 392228, Kurashiki-Shi
  - Investigational Site Number 392229, Matsuyama
  - Investigational Site Number 392230, Matsuyama
  - Investigational Site Number 392211, Mitaka-Shi
  - Investigational Site Number 392220, Nagoya
  - Investigational Site Number 392227, Nishinomiya-Shi
  - Investigational Site Number 392203, Ogawa-Machi, Hikigun
  - Investigational Site Number 392231, Okawa-Shi
  - Investigational Site Number 392224, Osaka
  - Investigational Site Number 392207, Shinjuku-Ku
  - Investigational Site Number 392219, Shizuoka
  - Investigational Site Number 392221, Takatsuki-Shi
  - Investigational Site Number 392202, Ushiku-Shi
  - Investigational Site Number 392213, Yokohama
  - Investigational Site Number 392214, Yokohama

REFERENCES:
- [Derived] Bolli GB, Wysham C, Fisher M, Chevalier S, Cali AMG, Leroy B, Riddle MC. A post-hoc pooled analysis to evaluate the risk of hypoglycaemia with insulin glargine 300 U/mL (Gla-300) versus 100 U/mL (Gla-100) over wider nocturnal windows in individuals with type 2 diabetes on a basal-only insulin regimen. Diabetes Obes Metab. 2019 Feb;21(2):402-407. doi: 10.1111/dom.13515. Epub 2018 Oct 2. PMID 30160030
- [Derived] Terauchi Y, Koyama M, Cheng X, Takahashi Y, Riddle MC, Bolli GB, Hirose T. New insulin glargine 300 U/ml versus glargine 100 U/ml in Japanese people with type 2 diabetes using basal insulin and oral antihyperglycaemic drugs: glucose control and hypoglycaemia in a randomized controlled trial (EDITION JP 2). Diabetes Obes Metab. 2016 Apr;18(4):366-74. doi: 10.1111/dom.12618. Epub 2016 Jan 21. PMID 26662838